CLINICAL TRIAL: NCT04529343
Title: Evaluation of the Effectiveness of Virtual Reality-Based Upper Extremity Rehabilitation in Patients With Cerebral Palsy
Brief Title: Virtual Reality Mediated Upper Extremity rehabilitationPatients With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ahmet Kivanc Menekseoglu, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/1442
Record Dates: First submitted 2020-08-18; First posted 2020-08-27 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Palsy; Upper Extremity Paresis
Keywords: virtual reality; rehabilitation; gamification
MeSH Terms: conditions — Cerebral Palsy; Paresis

STUDY DESIGN:
Intervention Model Description: The virtual reality group will be given upper extremity rehabilitation via virtual reality glasses (3 days a week for 6 weeks and 45 minutes each session) and upper extremity exercises 2 days a week, while the control group will only be given upper extremity exercises 2 days a week.
Who Masked: Outcomes Assessor
Masking Description: Assisting Hand Assessment was planned to be used in the evaluation of upper extremity functions as the primary outcome assessment tool. The person making this assessment will be blind to the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): To the virtual reality group; In addition to upper extremity exercises applied 2 days a week, upper extremity rehabilitation via virtual reality glasses will be performed 3 days a week for 6 weeks and each session will be 45 minutes.
  Interventions: Other: Virtual reality mediated upper extremity rehabilitation; Other: Classical exercise therapy for upper extremities
- Control Group (Active Comparator): Upper extremity exercises will be applied to the participants in the control group 2 days a week for 6 weeks.
  Interventions: Other: Classical exercise therapy for upper extremities

INTERVENTIONS:
Other: Virtual reality mediated upper extremity rehabilitation — Game-based exercise will be applied for different range of motion of the upper extremity. Gamified exercise program consisting of 4 different scenarios will be applied 3 days a week for 6 weeks to the patients in the virtual reality group. A session takes an average of 45 minutes.
  Games to be applied;
  1. Finger flexion-extension (10 minutes / session)
  2. Wrist flexion, extension, ulnar and radial deviation (10 minutes / session)
  3. Forearm pronation and supination (10 minutes / session)
  4. Elbow flexion-extension-shoulder internal and external rotation (15 minutes / session) will have scenarios controlled with. All patients participating in the study will receive exercise therapy in the form of upper extremity stretching, range of motion, and fine skill training 2 days a week for 6 weeks. Each session takes an average of 45 minutes.
  Arms: Virtual Reality Group
Other: Classical exercise therapy for upper extremities — All patients participating in the study will receive exercise therapy in the form of upper extremity stretching, range of motion, and fine skill training 2 days a week for 6 weeks. Each session takes an average of 45 minutes.

SUMMARY:
Cerebral palsy (CP) refers to a group of permanent disorders that occur in the brain of the fetus or infant, which are non-progressive, cause movement and posture disorder along with activity limitation.

The upper extremity is frequently affected in patients with CP. The prevalence of upper extremity involvement has been reported between 60-83% in different studies.

Virtual reality applications have been increasing recently in the field of neurological rehabilitation. In this study, researchers aimed to investigate the effectiveness of virtual reality-mediated upper extremity rehabilitation in patients with hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a group of permanent disorders of movement and posture development due to non-progressive damage to the developing fetal or infant brain, causing activity limitation. Motor disorders in CP are mostly accompanied by sensory and perceptual problems, cognitive disorders, communicative and perceptual problems, epilepsy and secondary musculoskeletal problems. CP is one of the most common causes of disability in childhood. Brain damage that causes CP can occur in the prenatal, perinatal or postnatal period. Accompanying epilepsy, cognitive disorders, learning impairment, communication problems, perception limitation, behavioral problems, visual disturbances, hearing disorders, oral motor function problems, dysphagia, constipation, gastroesophageal reflux disease, dental problems, urinary symptoms, osteoporosis can be seen in patients with CP.

Technologies that are developing in rehabilitation are increasingly being used. Among these technologies, the use of virtual reality by trained physiatrists and physiotherapists provides an environment where children with cerebral palsy can exercise. In addition to intense exercise, simultaneous visual and auditory feedback can be received. Virtual reality can also provide a comparison between the degree of movement children perform in the real world and the degree of movements they observe in the virtual environment. All these features make virtual reality a potentially viable tool for improving the motor skills of children with CP.

Virtual reality-based rehabilitation is an emerging treatment modality for the motor rehabilitation of children with cerebral palsy. Neuroplasticity studies have shown that neurological development is positively associated with active participation and motivation during virtual reality-based rehabilitation intervention. In addition to motivation, virtual therapy also improves neural reorganization that optimizes rehabilitation outcomes in children with cerebral palsy. The virtual scenario seems to encourage motor learning, the retention of learned skills, and the transfer of skills to real-world situations. In many studies, improvement in posture, balance, upper extremity functions, joint control and walking has been detected with virtual therapy. Increased 'biofeedbacks' in neuromotor rehabilitation allowed therapists to methodologically design and control their intervention strategies.

40 patients with a diagnosis of Cerebral Palsy who applied to the Pediatric Rehabilitation Unit of Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, who meet the inclusion criteria will be included in this randomized, controlled, single blind and prospectively planned study. At the beginning of the study, 40 hemiplegic CP patients who meet the inclusion criteria will be randomized into two groups according to the random order created by the computer program after being numbered according to the order of application to Istanbul University, Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Pediatric Rehabilitation Unit. Upper extremity rehabilitation (bimanually 3 days a week for 6 weeks and 45 minutes per session) and physiotherapy (TG: Treatment Group) will be given to the first group accompanied by virtual reality, and only physiotherapy (CG: Control Group) will be given to the second group.

When the power analysis was performed to calculate the number of patients and when the results obtained from other studies were taken into account, it was concluded that at least 18 patients should be included in each group to obtain 0.95 power at 95% confidence interval. Considering that few people will be excluded from the study during the study, it was found appropriate to include 20 patients in each group and to start the study with a total of 40 people. Before starting the study, the patients will be informed about the study and their consent will be obtained and demographic characteristics such as age, height and weight will be evaluated.

Participants and their parents will be informed in writing and verbally about the purpose, duration and method of application of the research, and the "Informed Consent Form" will be signed after their consent is obtained.

The study is planned to be carried out in a single center in the Department of Physical Medicine and Rehabilitation of Istanbul University Istanbul Medical Faculty.

The virtual reality technology to be used in the study has temporary side effects such as nausea, vomiting, and dizziness, and side effects to increase epileptic seizures. For this reason, patients with uncontrolled epileptic seizures were excluded from the study. If effects such as nausea, vomiting and dizziness develop during the intervention, the session will be terminated and symptomatic treatment will be given.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with hemiplegic CP by a specialist pediatric neurologist,
* Being between the ages of 5-12,
* Following the child's simple commands and participating in the given tasks,
* Being at the Gross Motor Function Classification System (KMFSS) Stage 1, 2 or 3,
* Being in Hand Skills Classification System (MACS) Stage 1, 2 or 3,
* Mild / moderate muscle tone; Modified Ashworth Scale level 1-2 and Tardieu Scale level 1-2,
* Parents agree to participate in the intensive treatment program and to cease all other upper extremity therapeutic interventions during the 3-month follow-up period.

Exclusion Criteria:

* Having uncontrollable epileptic seizures
* Significant contractures in the fingers, wrists, elbows and shoulders that prevent daily activities,
* Having serious vision and hearing problems,
* Cognitive impairments that prevent understanding and performing simple commands and tasks,
* Not being able to continue the treatment protocol due to the school program,
* Current or previous treatments that are not compatible with the treatment protocol of the study,
* Orthopedic surgery (tendon transfer / tendon lengthening) applied to the upper extremity,
* Receiving upper extremity treatment within the last 6 months (BTX-A or orthopedic interventions),
* Uncontrolled disease (endocrinological, cardiovascular, pulmonary, hematological, hepatic, renal), active systemic inflammatory disease and / or history of malignancy

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Assisting Hand Assessment (AHA) | 12 weeks
  AHA is a test that measures how patients with impaired upper extremity functions, such as hemiplegic CP or congenital brachial plexus injury, use the affected hand together with the healthy hand when playing with both hands. The AHA 5.0 version consists of 20 items that evaluate hand functions, and the raw score range is between 20 and 80 points. Higher scores indicate better hand function.

SECONDARY OUTCOMES:
Joint Range of Motion Measurement | 12 weeks
  Goniometric measurements of upper extremity range of motion will be done actively and passively.
Modified Ashworth Scale | 12 weeks
  Evaluation of upper extremity spasticity will be done with a modified Ashworth scale.The modified ashworth scale is scored between 0 and 4, with higher scores indicating severe spasticity.
Tardieu Scale | 12 weeks
  Evaluation of upper extremity spasticity will be done with a Tardieu scale. The Tardieu scale is scored between 0 and 5, with higher scores indicating severe spasticity.
ABILHAND-Kids | 12 weeks
  ABILHAND-Kids is a functional scale that is used to measure hand ability in patients, guiding the treatment planning of CP and similar childhood neurological diseases, determining targets. ABILHAND-Kids evaluates the hand functions of patients with 21 items, and each item is scored between 0-2 points. Higher scores indicate better hand function. (Minimum: 0, Maximum: 42 points)
QUEST | 12 weeks
  Upper extremity motion quality and hand skills of patients with CP were evaluated by QUEST.
  This test consists of 5 parts. In the test, each item is scored between 0 and 2, depending on whether it can perform the action or not. It has subtitles including independent movements, grasping, weight bearing, protective extension, hand function degree, spasticity rating and cooperation rating. Higher scores indicate better upper limb function. (Minimum: 0, Maximum: 100 points)
KINDL | 12 weeks
  KINDL is a questionnaire prepared in 1994 to evaluate the quality of life in the pediatric population and adolescents. There are various forms of the questionnaire for children of different age groups and families. The items in this test are scored between 1-5 points. Higher scores indicate better upper limb function. (Minimum: 0, Maximum: 100 points)

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Resa Aydın, Prof. Dr., Principal Investigator — Istanbul University Istanbul Medicine Faculty
Locations (1):
- Ahmet Kıvanç Menekşeoğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The patient data kept in the study will be shared with other researchers in case of a possible scientific publication. Personal data of the patients will not be shared, data of primary and secondary outcome criteria will be shared.

REFERENCES:
- [Result] Ravi DK, Kumar N, Singhi P. Effectiveness of virtual reality rehabilitation for children and adolescents with cerebral palsy: an updated evidence-based systematic review. Physiotherapy. 2017 Sep;103(3):245-258. doi: 10.1016/j.physio.2016.08.004. Epub 2016 Sep 27. PMID 28109566
- [Result] Cho C, Hwang W, Hwang S, Chung Y. Treadmill Training with Virtual Reality Improves Gait, Balance, and Muscle Strength in Children with Cerebral Palsy. Tohoku J Exp Med. 2016 Mar;238(3):213-8. doi: 10.1620/tjem.238.213. PMID 26947315
- [Result] Chen Y, Fanchiang HD, Howard A. Effectiveness of Virtual Reality in Children With Cerebral Palsy: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Phys Ther. 2018 Jan 1;98(1):63-77. doi: 10.1093/ptj/pzx107. PMID 29088476
- [Result] Ren Z, Wu J. The Effect of Virtual Reality Games on the Gross Motor Skills of Children with Cerebral Palsy: A Meta-Analysis of Randomized Controlled Trials. Int J Environ Res Public Health. 2019 Oct 14;16(20):3885. doi: 10.3390/ijerph16203885. PMID 31614990
- [Result] Hung YC, Gordon AM. Virtual reality training for children with unilateral cerebral palsy. Dev Med Child Neurol. 2018 Apr;60(4):334-335. doi: 10.1111/dmcn.13699. Epub 2018 Feb 14. No abstract available. PMID 29442357
- [Result] Ayed I, Ghazel A, Jaume-I-Capo A, Moya-Alcover G, Varona J, Martinez-Bueso P. Vision-based serious games and virtual reality systems for motor rehabilitation: A review geared toward a research methodology. Int J Med Inform. 2019 Nov;131:103909. doi: 10.1016/j.ijmedinf.2019.06.016. Epub 2019 Jul 10. PMID 31557701
- [Derived] Menekseoglu AK, Capan N, Arman S, Aydin AR. Effect of a Virtual Reality-Mediated Gamified Rehabilitation Program on Upper Limb Functions in Children With Hemiplegic Cerebral Palsy: A Prospective, Randomized Controlled Study. Am J Phys Med Rehabil. 2023 Mar 1;102(3):198-205. doi: 10.1097/PHM.0000000000002060. Epub 2022 Jun 9. PMID 35687751

DOCUMENTS (1):
  • Informed Consent Form (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT04529343/ICF_000.pdf